CLINICAL TRIAL: NCT00941031
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Regimen Finding Study of Subcutaneously Administered AIN457, Assessing Psoriasis Area and Severity Index (PASI) Response in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: AIN457 Regimen Finding Study in Patients With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2211; 2008-007525-39 (EudraCT Number)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Plaque-type Psoriasis
Keywords: Moderate to severe chronic plaque-type psoriasis; AIN457; dermatology
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Induction Single Dose (Experimental): Induction with single injection - "Single": secukinumab (AIN457) 150 mg s.c. administered at Week 1, Baseline through Week 12
  Interventions: Drug: AIN457
- Induction Monthly Dose (Experimental): Induction with monthly injections - "Monthly": secukinumab (AIN457) 150 mg s.c. administered at weeks 1, 5, 9, Baseline through Week 12
  Interventions: Drug: AIN457A
- Induction Early Loading Dose (Experimental): Early loading induction - "Early": secukinumab (AIN457) 150 mg s.c. administered at weeks 1, 2, 3, 5, Baseline through Week 12
  Interventions: Drug: AIN457A
- Placebo Dose (Placebo Comparator): Placebo administered at weeks 1, 2, 3, 5, 9, Baseline through Week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457
  Other Names: Secukinumab
  Arms: Induction Single Dose
Drug: AIN457A — Induction with monthly injections - "Monthly": secukinumab (AIN457) 150 mg s.c. administered at weeks 1, 5, 9
  Other Names: Secukinumab
  Arms: Induction Monthly Dose
Drug: AIN457A — Early loading induction - "Early": secukinumab (AIN457) 150 mg s.c. administered at weeks 1, 2, 3, 5
  Other Names: Secukinumab
  Arms: Induction Early Loading Dose
Drug: Placebo — Placebo - "Placebo": Placebo administered at weeks 1, 2, 3, 5, 9
  Arms: Placebo Dose

SUMMARY:
The purpose of the study is to determine whether, in patients with moderate to severe plaque-type psoriasis, AIN457 administered subcutaneously reduces the severity of psoriasis symptoms and the extent to which the patient's body area is affected by the disease (compared to placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age at time of consent
* Chronic plaque-type psoriasis diagnosed for at least 6 months at time of randomization
* At time of randomization, moderate to severe psoriasis as defined by:

  * PASI score of 12 or greater and
  * IGA score of 3 or greater and
  * Body Surface Area (BSA) affected by plaque-type psoriasis of 10 % or greater
* At screening and randomization, chronic plaque-type psoriasis considered inadequately controlled by:

  * topical treatment and/or
  * phototherapy and/or
  * previous systemic therapy

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from entry into the study:
* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at screening or randomization
* Drug-induced psoriasis (i.e. new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) and randomization
* Ongoing use of prohibited psoriasis treatments (e.g., topical or systemic corticosteroids, UV therapy) at randomization. Washout periods detailed in the study protocol have to be adhered to
* Ongoing use of other prohibited treatments at randomization. Washout periods detailed in the study protocol have to be adhered to. All prior concomitant medications must be on a stable dose for at least four weeks before study drug administration
* Known immunosuppression (e.g., AIDS) at screening and / or randomization
* History or evidence of active tuberculosis at screening. All patients will be tested for tuberculosis status using a blood test (QuantiFERON®-TB Gold In-Tube). Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment has been initiated according to local regulations.
* Active systemic infections (other than common cold) during the two weeks before randomization (e.g., hepatitis)
* At screening, history or symptoms of malignancy of any organ system (other than history of basal cell carcinoma and / or up to three squamous cell carcinomas of the skin, if successful treatment has been performed, with no signs of recurrence; actinic keratoses, if present at screening, should be treated according to standard therapy before randomization), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* History of congestive heart failure (NYHA functional classification ≥III) at screening and / or randomization
* History of severe hypersensitivity to any human or humanized biological agents (antibody or soluble receptor) at screening and / or randomization
* Any severe, progressive or uncontrolled medical condition at randomization that in the judgment of the investigator prevents the patient from participating in the study
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (28):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Newnan, Georgia
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Clinton Twp., Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Lynchburg, Virginia
- France (2):
  - Novartis Investigative Site, Toulouse, France
  - Novartis Investigative Site, Nice
- Germany (14):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Kopavogur, Iceland
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Chitose, Hokkaido
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Norway (3):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo

REFERENCES:
- [Derived] Paul C, Reich K, Gottlieb AB, Mrowietz U, Philipp S, Nakayama J, Harfst E, Guettner A, Papavassilis C; CAIN457A2211 study group. Secukinumab improves hand, foot and nail lesions in moderate-to-severe plaque psoriasis: subanalysis of a randomized, double-blind, placebo-controlled, regimen-finding phase 2 trial. J Eur Acad Dermatol Venereol. 2014 Dec;28(12):1670-5. doi: 10.1111/jdv.12359. Epub 2014 Jan 7. PMID 24393602

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Early Loading: Early loading induction - "Early": secukinumab (AIN457) 150 mg s.c. administered at weeks 1, 2, 3, 5, Baseline through Week 12
- Fixed Interval: Fixed-time interval regimen - "FI": secukinumab (AIN457) 150 mg s.c. administered at Week 13 and at Week 25 and placebo at regular scheduled visit at which a start of relapse was observed, Week 21 to Week 29
- Start of Relapse: Treatment at start of relapse regimen - "SR": Placebo administered at Week 13 and possibly at Week 25 if no start of relapse observed, and secukinumab (AIN457) 150 mg s.c. administered at regular scheduled visit at which a start of relapse was observed, Week 21 to Week 29
- Open Label: Non responders and partial responders at Week 13 and patients who experienced 2 consecutive relapses at scheduled visits from Week 13 onwards were eligible to enter the Open Label phase - "OL": secukinumab (AIN457) 150 mg s.c. administered every 4 weeks.21 to Week 29
Period: Induction Period
Arm/Group | Induction Single Dose | Induction Monthly Dose | Induction Early Loading | Placebo Dose | Fixed Interval | Start of Relapse | Open Label
Started | 66 | 138 | 133 | 67 | 0 | 0 | 0
Completed | 61 | 134 | 127 | 58 | 0 | 0 | 0
Not Completed | 5 | 4 | 6 | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 2 | 0 | 0 | 0
Not completed — Adminstative Problems | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 3 | 2 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Induction Single Dose | Induction Monthly Dose | Induction Early Loading | Placebo Dose | Fixed Interval | Start of Relapse | Open Label
Started | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Non Responders treated with an open label regimen.) | 65 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 67 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 247 (Non Responders treated with an open label regimen.)
Completed | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Responders at week 13 were re randomized to one of the maintenance treatment arms in a ratio of 1:1) | 0 (Non Responders treated with an open label regimen.) | 56 | 61 | 204
Not Completed | 0 | 0 | 0 | 0 | 9 | 6 | 43
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 6 | 2 | 13
Not completed — Administrative Problems | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 2 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Induction Single Dose: Baseline through Week 12
- Total: Total of all reporting groups
Arm/Group | Induction Single Dose | Induction Monthly Dose | Induction Early Loading Dose | Placebo | Total
Number analyzed (Participants) | 66 | 138 | 133 | 67 | 404
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (11.32) | 44.2 (12.96) | 44.5 (12.45) | 44.2 (12.59) | 44.1 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 34 | 28 | 23 | 98
  Male | 53 | 104 | 105 | 44 | 306
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 17 | 14 | 8 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 59 | 120 | 118 | 56 | 353
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Three Induction Regimens of AIN457 Administered Subcutaneously in Patients With Moderate to Severe Chronic Plaque-type Psoriasis With Respect to PASI 75 Achievement After 12 Weeks of Treatment, Compared to Placebo.
Description: Number (%) of patients achieving PASI 50, PASI 75, PASI 90, by visit and induction treatment
Time Frame: 13 weeks
Population: (Full analysis set, LOCF) Number (%) of patients achieving PASI 50, PASI 75, PASI 90, by visit and induction treatment
Measure: Number; unit: Participants achieving goal
Arm/Group | Induction Single Dose | Induction Monthly Dose | Induction Early Loading Dose | Placebo Dose
Number analyzed (Participants) | 66 | 138 | 132 | 66
Participants achieving goal
  PASI 50 | 18 | 83 | 101 | 7
  PASI 75 | 7 | 58 | 72 | 1
  PASI 90 | 2 | 24 | 42 | 1

2. Secondary Outcome: The Efficacy of Two Maintenance Regimens of AIN457 With Respect to PASI 75 Achievement at Least Once From Week 21 to 29
Time Frame: week 21 to 29
Population: (Full analysis set, LOCF)
Measure: Number; unit: Participants achieving goal
Groups:
- Maintenance Fixed Interval: Fixed-time interval regimen - "FI": secukinumab (AIN457) 150 mg s.c. administered at Week 13 and at Week 25 and placebo at regular scheduled visit at which a start of relapse was observed, Week 21 to Week 29
- Maintenance Start of Relapse: Treatment at start of relapse regimen - "SR": Placebo administered at Week 13 and possibly at Week 25 if no start of relapse observed, and secukinumab (AIN457) 150 mg s.c. administered at regular scheduled visit at which a start of relapse was observed, Week 21 to Week 29
- Maintenance Open Label: Non responders and partial responders at Week 13 and patients who experienced 2 consecutive relapses at scheduled visits from Week 13 onwards were eligible to enter the Open Label phase - "OL": secukinumab (AIN457) 150 mg s.c. administered every 4 weeks.21 to Week 29
Arm/Group | Maintenance Fixed Interval | Maintenance Start of Relapse | Maintenance Open Label
Number analyzed (Participants) | 65 | 67 | 247
Participants achieving goal
  PASI 50 | 64 | 60 | 200
  PASI 75 | 55 | 45 | 114
  PASI 90 | 38 | 14 | 53

3. Secondary Outcome: The Efficacy of Three Induction Regimens of AIN457 Administered Subcutaneously With Respect Participants Who Reported Either an IGA 0 or 1 After 12 Weeks of Treatment, Compared to Placebo
Description: The investigator's global assessment (IGA) was used to evaluate overall psoriatic disease, with scores ranging from 0 (clear) to 5 (very severe disease). Treatment success was defined as patients who achieved IGA 0 or 1 and improvement of at least 2 points on the IGA scale compared to baseline. The IGA rating score for involvement of hands and feet ranged from 0 (clear) to 4 (severe).
Time Frame: 13 weeks
Population: Full analysis set
Measure: Number; unit: Participants achieving goal
Arm/Group | Induction Single Dose | Induction Monthly Dose | Induction Early Loading Dose | Placebo Dose
Number analyzed (Participants) | 66 | 137 | 132 | 66
Participants achieving goal
  0=clear | 0 | 2 | 17 | 1
  1= almost clear | 3 | 29 | 32 | 0
  2= mild disease | 17 | 42 | 38 | 3
  3= moderate disease | 28 | 44 | 33 | 26
  4=severe disease | 15 | 18 | 12 | 29
  5= very serious disease | 3 | 2 | 0 | 7

ADVERSE EVENTS:
Groups:
- INDUCTION: Single: INDUCTION: Early loading induction - 'Early'
- INDUCTION: Monthly: INDUCTION: with monthly injections - 'Monthly'
- INDUCTION: Early: INDUCTION: with single injection - 'Single'
- INDUCTION: Placebo: INDUCTION: Placebo - 'Placebo'
- MAINTENANCE: Fixed Interval: MAINTENANCE: Fixed-time interval regimen - 'FI'
- MAINTENANCE: Start of Relapse: MAINTENANCE: Treatment at start of relapse regimen - 'SR'
- MAINTENANCE: Open Label: MAINTENANCE: Open label Non responders and partial responders at Week 13 and patients who experienced 2 consecutive relapses at scheduled visits from Week 13 onwards were eligible to enter the Open Label phase - "OL": secukinumab (AIN457) 150 mg s.c. administered every 4 weeks.
- FOLLOW-UP: Fixed Interval: FOLLOW-UP: Fixed-time interval regimen - 'FI'
- FOLLOW-UP: Start of Relapse: FOLLOW-UP: Treatment at start of relapse regimen - 'SR'
- FOLLOW-UP: Open Label: FOLLOW-UP: Open label
Arm/Group | INDUCTION: Single | INDUCTION: Monthly | INDUCTION: Early | INDUCTION: Placebo | MAINTENANCE: Fixed Interval | MAINTENANCE: Start of Relapse | MAINTENANCE: Open Label | FOLLOW-UP: Fixed Interval | FOLLOW-UP: Start of Relapse | FOLLOW-UP: Open Label
Serious Adverse Events (participants affected / at risk) | 3/66 | 3/138 | 6/133 | 1/67 | 4/65 | 2/67 | 12/247 | 0/17 | 0/15 | 5/72
Other Adverse Events (participants affected / at risk) | 23/66 | 53/138 | 46/133 | 29/67 | 16/65 | 16/67 | 83/247 | 3/17 | 4/15 | 5/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION: Single (N=66) | INDUCTION: Monthly (N=138) | INDUCTION: Early (N=133) | INDUCTION: Placebo (N=67) | MAINTENANCE: Fixed Interval (N=65) | MAINTENANCE: Start of Relapse (N=67) | MAINTENANCE: Open Label (N=247) | FOLLOW-UP: Fixed Interval (N=17) | FOLLOW-UP: Start of Relapse (N=15) | FOLLOW-UP: Open Label (N=72)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION: Single (N=66) | INDUCTION: Monthly (N=138) | INDUCTION: Early (N=133) | INDUCTION: Placebo (N=67) | MAINTENANCE: Fixed Interval (N=65) | MAINTENANCE: Start of Relapse (N=67) | MAINTENANCE: Open Label (N=247) | FOLLOW-UP: Fixed Interval (N=17) | FOLLOW-UP: Start of Relapse (N=15) | FOLLOW-UP: Open Label (N=72)
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 31 | 30 | 12 | 6 | 5 | 35 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 2 | 6 | 2 | 0 | 17 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 0 | 0 | 1 | 1 | 9 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 8 | 11 | 3 | 3 | 1 | 13 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 4 | 0 | 0 | 8 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 7 | 4 | 6 | 4 | 6 | 16 | 2 | 1 | 1
Hypertension (Vascular disorders) | 3 | 1 | 2 | 1 | 2 | 5 | 5 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial